CLINICAL TRIAL: NCT01641471
Title: Prospective Evaluation of Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Relief Following Total Knee Arthroplasty (TKA)
Brief Title: Evaluation of Electrical Nerve Stimulation (TENS) Therapy for Pain Relief Following Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Principal Investigator, Wael Barsoum, MD, Chairman of Surgical Operations, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCF 12-476
Record Dates: First submitted 2012-06-19; First posted 2012-07-16 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Knee; Arthritis; Pain
Keywords: Total Knee Arthroplasty (TKA); Transcutaneous Electrical Nerve Stimulation (TENS); Pain; Function; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TENS (Experimental): Active TENS (EMPI Select TENS) in combination with a femoral nerve catheter. Patients will begin using the TENS unit immediately following surgery and continuing throughout the 6 weeks postoperatively.
  Interventions: Device: EMPI Select TENS
- Placebo TENS (Placebo Comparator): Placebo TENS (Placebo EMPI Select TENS) in combination with a femoral nerve catheter. Patients will begin using a sham TENS unit (appears identical to Active TENS unit, yet is created to deliver low-level, non-therapeutic electrical stimulation) immediately following surgery and continuing throughout the 6 weeks postoperatively.
  Interventions: Device: Placebo EMPI Select TENS

INTERVENTIONS:
Device: EMPI Select TENS — The unit is capable of 0-60 milliamps of output current.
  Arms: Active TENS
Device: Placebo EMPI Select TENS — The sham unit appears identical to the Active TENS unit, yet is created to deliver low-level, non-therapeutic electrical stimulation.
  Arms: Placebo TENS

SUMMARY:
Evaluation of Electrical Nerve Stimulation (TENS) Therapy for Pain Relieft Following Total Knee Arrhtoplasty (TKA)

DETAILED DESCRIPTION:
A prospective, randomized postmarket trial to assess the efficacy of the Select TENS™ Pain Management System, a transcutaneous electrical nerve stimulation (TENS) device, for reducing pain and narcotics requirement in patients managed with a total knee arthroplasty (TKA). This will be a placebo-controlled study involving 116 patients undergoing primary unilateral TKA procedures; 58 patients will be randomly selected to be treated postoperatively with an active TENS unit and the other 58 patients will be randomly selected to be treated with the placebo TENS unit (control group). Patients will be enrolled at two sites within the Cleveland Clinic Health System (Main Campus and Lutheran Hospital). Both treatment and control groups will receive a femoral nerve catheter, standard during a primary TKA. It is hypothesized that TENS (in combination with a femoral nerve catheter) can reduce narcotic usage, reduce pain, and allow for a quicker return to function following TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total knee arthroplasty
* Patients who are between the ages of 18-85 years
* Patient has signed informed consent

Exclusion Criteria:

* Patients who live >100 miles from the Cleveland Clinic main campus (9500 Euclid Ave., Cleveland, OH 44195)
* Patients who will not receive a femoral nerve catheter for surgery
* Patients who are not planned to be discharged directly home following surgery
* Patients who have used a TENS device in the past
* Preoperative daily use of narcotics (i.e., high tolerance)
* Already enrolled in another research study, including the present study for contralateral knee
* Patients with a history of epilepsy
* Patients with a cardiac pacemaker
* Patients who are a risk for poor compliance or have a poor understanding of the use of the TENS device
* Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornell PE, Lopez AL, Malofsky H. Pain reduction with transcutaneous electrical nerve stimulation after foot surgery. J Foot Surg. 1984 Jul-Aug;23(4):326-33. PMID 6332127
- [Background] Arvidsson I, Eriksson E. Postoperative TENS pain relief after knee surgery: objective evaluation. Orthopedics. 1986 Oct;9(10):1346-51. doi: 10.3928/0147-7447-19861001-06. PMID 3490659
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] Breit R, Van der Wall H. Transcutaneous electrical nerve stimulation for postoperative pain relief after total knee arthroplasty. J Arthroplasty. 2004 Jan;19(1):45-8. doi: 10.1016/s0883-5403(03)00458-3. PMID 14716650

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TENS: Active TENS in combination with a femoral nerve catheter. Patients will begin using the TENS unit immediately following surgery and continuing throughout the 6 weeks postoperatively.
  EMPI Select TENS: The unit is capable of 0-60 milliamps of output current. The 4 electrodes will be focused on the posterior aspect of the knee during the immediate postoperative period and lasting through discharge from the hospital. Once the patient is discharged, he/she will be instructed to use the device as he/she would like, whether it is a continuation of the posterior placement of the electrodes, or a more traditional anterior criss-cross positioning. Patients will be instructed to use the device for 2 hours on, followed by 30 minutes off, as needed. Amount of TENS usage and average intensity used will be recorded. An assessment of blinding will be conducted at the conclusion of the study by asking patients what treatment arm they think that they received.
- Placebo TENS: Placebo TENS in combination with a femoral nerve catheter. Patients will begin using a sham TENS unit (appears identical to Active TENS unit, yet is created to deliver low-level, non-therapeutic electrical stimulation) immediately following surgery and continuing throughout the 6 weeks postoperatively.
  Placebo EMPI Select TENS: Sham unit appears identical to the Active TENS unit, yet is created to deliver low-level, non-therapeutic electrical stimulation (even though screen shows 0-60 milliamps of output current). The 4 electrodes will be focused on the posterior aspect of the knee during immediate postoperative period and lasting through discharge from the hospital. Once patient is discharged, he/she will be instructed to use the device as he/she would like, whether it is a continuation of the posterior placement of the electrodes, or a more traditional anterior criss-cross positioning. Patients will be instructed to use the device for 2 hours on, followed by 30 minutes
Period: Overall Study
Arm/Group | Active TENS | Placebo TENS
Started | 58 | 58
Completed | 35 | 31
Not Completed | 23 | 27
Not completed — Withdrawal by Subject | 19 | 19
Not completed — Lost to Follow-up | 2 | 4
Not completed — Protocol Violation | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TENS | Placebo TENS | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (3.7) | 60.3 (7.7) | 62.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Usage
Description: Morphine Equivalent dose, mg/kg
Time Frame: Through 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 35 | 31
morphine equivalents | 997.7 (1124.9) | 1025.8 (1053.6)

2. Secondary Outcome: Visual Analog Pain Score (VAS)
Description: Pain VAS is a continuous scale comprised of a vertical line, 10 centimeters in length, with each centimeter marked by its' corresponding whole number (1, 2, 3, etc.). It ranges from 0 to 10, with 0 being no pain and 10 being maximum pain.
Time Frame: 6 weeks (+/- 3 days) postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 35 | 31
units on a scale | 1.57 (1.35) | 1.54 (1.52)

3. Secondary Outcome: Functional Assessments
Description: Timed up and go (TUG) test. These methods follows those published by Podsiadlo and Richardson, JAGS 1991; 39:142-148, in which the patient is observed and timed while he/she rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.
Time Frame: 6 weeks (+/- 3 days) postoperative
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 35 | 31
seconds | 9.31 (2.67) | 10.39 (4.29)

4. Secondary Outcome: General Health Outcome - SF-12 Physical Component Summary
Description: Physical Component Score. Physical Component Score (PCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. PCS provides emphasis on questions about general health, physical functioning and role playing and bodily pain. PCS is standardized using a z-score transformation and normed to a US population (Based on a 1990 norm) of a score of 50.0 and a standard deviation of 10.0. Normalized scores reported.
Time Frame: 6 weeks (+/- 3 days) postoperative
Measure: Mean (Standard Deviation); unit: z-scale
Arm/Group | Active TENS | Placebo TENS
Number analyzed (Participants) | 35 | 31
z-scale | 33.57 (7.02) | 31.78 (7.07)

ADVERSE EVENTS:
Arm/Group | Active TENS | Placebo TENS
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/31
Other Adverse Events (participants affected / at risk) | 10/35 | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=35) | Placebo TENS (N=31)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TENS (N=35) | Placebo TENS (N=31)
Blisters (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intraoperative MCL tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Postoperative ligament tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No